CLINICAL TRIAL: NCT04457765
Title: Povidine-Iodine Effect on Nasal Mucosa Cilia in Rhinoplasty Patients
Brief Title: Betadine Effect on Nasal Mucosa Cilia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The IRB did not approve the study to be conducted at the home institution.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-40432
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Rhinoplasty
Keywords: Septorhioplasty; Povidine-Iodine (PVP-I); Betadine; Nasal mucosa cilia (NMC); Saccharin transit time (STT)
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- group 1 (Experimental): All participants will have PVP-I at 1.25% administered as an intranasal topical preparation prior undergoing rhinoplasty
  Interventions: Drug: Povidone-Iodine (PVP-I)

INTERVENTIONS:
Drug: Povidone-Iodine (PVP-I) — 1.25% Povidone-Iodine (PVP-I) (also known as betadine) to be used pre-procedure in the operating room via irrigation into the nasal cavity to act as viricidal preparation for the procedure. 240mL of 1.25% PVP-I will be distributed evenly among the right and left nasal cavities using a a 70mL syringe.
  Other Names: Betadine

SUMMARY:
The goal of the proposed study is to identify PVP-I at 1.25% as an appropriate intranasal topical preparation for patients undergoing rhinoplasty with no effect on the nasal mucosa cilia (NMC) or olfaction using the saccharin transit time (STT) test as a method for evaluating NMC function. PVP-I has been shown to be viricidal in the upper aerodigestive tract. This study is highly-relevant, as protection for individuals with a high risk of exposure to respiratory pathogens has become increasingly important in the setting of recent viral epidemics such as SARS-CoV-2. Septorhinoplasty is commonly performed throughout the world and there is a paucity of standardized testing in surgical facilities. Much of our understanding of the current COVID-19 pandemic is extrapolated from MERS and SARS data. It is our hope that this study's relevance for the current pandemic remains so in the unfortunate event of another pandemic in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Boston Medical Center undergoing septorhinoplasty, without inferior turbinate reduction
* Normal range baseline saccharin transit time (STT)
* SARS-CoV-2 Testing Negative at the time of the procedure o Per institution guidelines, patients scheduled for surgery undergo a preoperative nasopharyngeal test within 24 hours of their procedure - per institution protocols.

Exclusion Criteria:

* Known history of:

  * thyroid dysfunction
  * renal disease
  * autoimmune disease affecting the upper airway
  * immunocompromised
  * pregnant, breastfeeding
* Patients determined to have dysfunctional nasal mucosa cilia (NMC) function based on a STT time of ≥30 minutes
* Patients with a contraindication to Povidone-iodine (PVP-I) including history of allergy/anaphylaxis to PVP-I, labile thyroid disease, history of contact dermatitis, active radioiodine therapy, pregnancy/nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Preoperative nasal mucosa cilia (NMC) function | baseline
  NMC will be assessed with the saccharin transit time (STT) test. This test is done by the examiner inserting sodium saccharin particle on the upper surface of the inferior nasal turbinate.The patient is instructed to swallow once every minute and notify the examiner when they notice a sweet taste. The distance from the start of the mucociliary membrane to far wall of pharynx is measured with a probe. From this measurement, the mean velocity is calculated compared to the total time from the start of the test. Dysfunction is defined as a STT >30.
Postoperative nasal mucosa cilia (NMC) function | 5 weeks
  NMC will be assessed with the saccharin transit time (STT) test. This test is done by the examiner inserting sodium saccharin particle on the upper surface of the inferior nasal turbinate.The patient is instructed to swallow once every minute and notify the examiner when they notice a sweet taste. The distance from the start of the mucociliary membrane to far wall of pharynx is measured with a probe. From this measurement, the mean velocity is calculated compared to the total time from the start of the test. Dysfunction is defined as a STT >30.

SECONDARY OUTCOMES:
Change in self reported symptoms of nasal blockage or obstruction | baseline, 5 weeks
  Nasal symptoms will be assessed with the NOSE (Nasal Obstruction Symptom Evaluation) Tool. NOSE has 5 questions and response options for each range from 0 to 4 where 0= Not a problem, 1= Mild problem, 2= Moderate problem, 3= Significant problem, 4= Severe problem. The response value for each question is multiplied by 5 so overall NOSE scores can range from 0 to 100 and are interpreted as-- 0: Nothing to worry about; 5 - 25: Mild obstruction; 26 - 50: Moderate obstruction; 51 - 75: Significant obstruction; 76 - 100: Severe obstruction.
Change in olfactory function | baseline, 5 weeks
  The participant will be instructed to sniff repetitively and to tell when an odor is detected, identifying the odor if recognized. The test odor up to within 30 cm or less of the nose.
Change in quality of life based on sino-nasal symptoms | baseline, 5 weeks
  Participants' quality of life will be assessed using the Sino-nasal Outcome Test (SNOT-22). This is a self administered questionnaire with 22 items. Each items is answered by selecting one of 6 categories where 0 = No problem, 1 = Very Mild problem, 2 = Mild or slight problem, 3 = Moderate problem, 4 = Severe problem, 5 = Problem as bad as it can be. Scores can range from 0 to 110. A score of 7 or below is considered 'normal' scores 8 or above suggests that sino-nasal symptoms are affecting participants' quality of life.
Preoperative clinical examination of nasal mucosa | baseline
  A through preoperative clinical examination of each participant will be done and findings documented.
Post operative clinical examination of nasal mucosa | 5 weeks
  A through postoperative clinical examination of each participant will be done and findings documented.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ezzat, MD, Study Chair — Boston Medical Center; Jennifer Shehan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No